CLINICAL TRIAL: NCT06762444
Title: Bump the Lump: Creation and Validation of Speech Language Pathology Intervention for the Treatment of Globus Pharyngeus
Brief Title: Bump the Lump - Intervention for the Treatment of Globus Pharyngeus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00103445
Record Dates: First submitted 2024-12-30; First posted 2025-01-07 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Globus Pharyngeus
Keywords: Speech-language pathologist; laryngeal hygiene; voice therapy techniques
MeSH Terms: conditions — Globus Sensation | interventions — Complement C4a; Clinical Protocols

STUDY DESIGN:
Intervention Model Description: The Speech-language pathologist (SLP) intervention protocol consists of six components, all of which will be implemented by the treating speech-language pathologist
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- The SLP intervention protocol (Experimental): The SLP intervention protocol consists of six components, all of which will be implemented by the treating speech-language pathologist
  Interventions: Behavioral: Speech-language pathologist (SLP) protocol

INTERVENTIONS:
Behavioral: Speech-language pathologist (SLP) protocol — The SLP intervention protocol consists of six components, all of which will be implemented by the treating speech-language pathologist

SUMMARY:
To develop a standardized speech-language pathology treatment protocol to systematically address Globus pharyngeus (GP) as a proof of concept

DETAILED DESCRIPTION:
Globus pharyngeus (GP), often described as a persistent lump or tightness in the throat, accounting for 4% of new referrals to Ear, Nose, and Throat (ENT) clinics. This condition is reported in the literature in up to 46% of healthy individuals and has been shown to significantly impact patients' quality of life. The key diagnostic criteria for GP include at least 12 weeks duration of symptoms without dysphagia or gastroesophageal reflux as the causative symptom, and in the absence of major esophageal motor disorders. While the exact etiology of GP remains elusive, research suggests a multifactorial nature involving physical, psychological, and functional components. Behavioral therapy with a Speech-language pathologist is often recommended as a treatment option for patients with GP. A review of the literature examining SLP interventions for GP shows that SLP treatments lack standardization, leading to inconsistency and limited efficacy across therapeutic interventions. Therefore, there is an urgent need to further investigate behavioral interventions for GP and develop a standardized treatment protocol to address the condition systematically.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer adult patients (age 18 and over) evaluated at the Atrium Health Wake Forest Baptist Center for Voice and Swallowing Disorders who report a complaint of globus pharyngeus

Exclusion Criteria:

* Patients diagnosed with a swallowing disorder will be excluded from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Laryngopharyngeal Measure of Perceived Sensation (LUMP) | Year 1
  Laryngopharyngeal Measure of Perceived Sensation (LUMP) to assess GP symptom severity - The Laryngopharyngeal Measure of Perceived Sensation (LUMP) scoring system is a patient-reported questionnaire used to assess the severity of throat sensations like globus sensation (lump in the throat) - where each item on the scale is rated 0 (never) to 4 (always), with a higher score indicating greater symptom severity - A LUMP score greater than or equal to 3 should be considered abnormal and warrants additional attention.
Eating Assessment Tool-10 (EAT-10) | Year 1
  Eating Assessment Tool-10 (EAT-10) to assess for dysphagia complaints - The Eating Assessment Tool (EAT-10) is increasingly used to screen for self-perceived oropharyngeal dysphagia (OD) in community-dwelling elders. A summated EAT-10 total score ranges from 0 to 40, with a score ≥ 3 is abnormal
Voice Handicap Index-10 (VHI-10) | Year 1
  Voice Handicap Index-10 (VHI-10) to measure voice-related quality of life - The Voice Handicap Index-10 (VHI-10) is a patient-reported outcome measure that scores voice-related handicap on a scale of 0-40:
  Normal or nearly normal: Scores of 0-10 Abnormal: Scores above 11 Greater handicap: Higher scores indicate a greater voice-related handicap
Generalized Anxiety Disorder-7 (GAD-7) | Year 1
  Generalized Anxiety Disorder-7 (GAD-7) to assess for anxiety - The Generalized Anxiety Disorder 7-item (GAD-7) is a self-report scale that assesses anxiety and worry symptoms. The GAD-7 score is calculated by adding up the scores for each of the seven items, with scores ranging from 0 to 21 - Score 0-4: Minimal Anxiety. Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety
Numeric Rating Scale for throat pain | Year 1
  0-10 Numeric Rating Scale for throat pain to assess for throat pain - a scale from 0 to 10, where "0" represents "no throat pain" and "10" represents "the worst throat pain imaginable

CONTACTS AND LOCATIONS:
Overall Officials: Lyndsay Madden, DO, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No